CLINICAL TRIAL: NCT05304195
Title: Exploration of Glucocerebrosidase Activity to Identify a Subpopulation Eligible for a Therapeutic Trial in Dementia With Lewy Bodies
Brief Title: Exploration of GCase Activity to Identify a Subpopulation Eligible for a Therapeutic Trial in Dementia With Lewy Bodies
Acronym: EGELY
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201175; 2021-A02345-36 (Other: IDRCB)
Record Dates: First submitted 2022-01-27; First posted 2022-03-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Dementia With Lewy Bodies
Keywords: Glucocerebrosidase; GBA gene
MeSH Terms: conditions — Lewy Body Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — GBA gene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DLB patients: Dementia with lewy bodies according to the revised criteria of Mc Keith 2017
  Interventions: Diagnostic Test: Glucocerebrosidase; Genetic: GBA gene; Diagnostic Test: Macrophage biomarkers
- Control: Absence of cognitive impairment and clinical element for a neurodegenerative disease
  Interventions: Diagnostic Test: Glucocerebrosidase; Genetic: GBA gene; Diagnostic Test: Macrophage biomarkers

INTERVENTIONS:
Diagnostic Test: Glucocerebrosidase — Blood sample (10ml) for GCase activity
Genetic: GBA gene — Blood sample (10ml) for variants or mutations of the GBA gene
Diagnostic Test: Macrophage biomarkers — Blood sample (20ml) for macrophage biomarkers

SUMMARY:
This research focuses on the activity of an enzymatic protein: glucocerebrosidase, in dementia with lewy bodies (DLB). Indeed, the mutation of the GBA gene responsible for a decrease in the activity of glucocerebrosidase is the most frequent known genetic risk factor in DLB. However, mutations of the GBA gene are known in another pathology, Gaucher disease, in which treatments have been developed.

The objective of this research is to determine if glucocerebrosidase activity is decreased in DLB. This hypothesis could open up a therapeutic perspective, with treatments already used in Gaucher disease.

DETAILED DESCRIPTION:
Population: 118 patients and 118 control subjects Act of research: blood test

Objectifs :

* Comparison of glucocerebrosidase activity between patients and controls
* Search for variants or mutations of the GBA gene and correlation with glucocerebrosidase activity
* Correlation between clinical characteristics (UPDRS motor scale, MMSE cognitive scale) and GCase activity in patients
* Identification of macrophage abnormalities and the impact of treatments targeting the GBA pathway on the deregulation of biomarkers in patient macrophages.

ELIGIBILITY:
Inclusion Criteria for patients :

* Male or female aged ≥ 50 years old
* Presence of an accompanying person
* Dementia with lewy bodies according to the revised criteria of Mc Keith 2017

Inclusion Criteria for controls:

* Male or female aged ≥ 50 years old
* Absence of cognitive impairment and clinical element for a neurodegenerative disease

Exclusion Criteria for patients:

* Other neurodegenerative disease
* Gaucher disease

Exclusion Criteria for controls:

* Neurodegenerative disease
* Cognitive impairment of all causes

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 118 patients and 118 control subjects Patients and controls (often an accompanying person) will be selected during a routine visit for the patient's DLB
Sampling Method: Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
GCase activity in patients and control by fluorometry | through study competion, an average of 1 year
  difference in measurement of glucocerebrosidase enzyme activity (by fluorometry method) between DLB patients and control subjects.

SECONDARY OUTCOMES:
GBA gene and GCase activity | through study competion, an average of 1 year
  correlation between the presence of GBA gene mutation and the measurement of glucocerebrosidase enzymatic activity
MMSE score and GCase activity | through study competion, an average of 1 year
  correlation between the measurement of glucocerebrosidase enzymatic activity and MMSE score (Mini-Mental State Examination from 0-severe to 30-normal) of DLB patients
motor sub-score of UPDRS score and GCase activity | through study competion, an average of 1 year
  correlation between the measurement of glucocerebrosidase enzymatic activity and motor sub-score of UPDRS score (motor sub-score of Unified Parkinson Disease Rating Scale from) of DLB patients The score is between 0 and 55. The score increases proportionally to the severity of the extrapyramidal syndrome.
GBA gene and macrophage abnormalities | through study competion, an average of 1 year
  Correlation between the presence of a GBA gene mutation and abnormal macrophage activation reflecting a specific inflammatory profile and biomarker variation.
Treatment and macrophage biomarkers | through study competion, an average of 1 year
  Identification of the impact of treatments targeting the GBA pathway on the deregulation of biomarkers in macrophages.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de neurologie Cognitive, Paris, France, France

IPD SHARING:
Plan to Share IPD: No